CLINICAL TRIAL: NCT05013203
Title: Next Generation Sequencing for the Detection of Clinical and Subclinical Infection in Patient Undergoing Spine Surgery
Brief Title: NGS for Spine Surgery Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Other Study IDs: CKEP21d.121
Record Dates: First submitted 2021-08-13; First posted 2021-08-19 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Spine Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Aseptic (uninfected) Revision Spine Surgery: Aseptic revision for indications including but not limited to hardware failure, adjacent segment pathology, radiculopathy, instability, cord compression.
  Interventions: Diagnostic Test: Tissue culture; Diagnostic Test: Next Generation Sequencing
- Spine Surgery for Degenerative Disease: Primary degenerative pathology surgery where a disc sample is extracted to enable spinal decompression or fusion. The potential primary surgeries include but are not limited to microdiscectomy, laminectomy, and lumbar and cervical fusion
  Interventions: Diagnostic Test: Tissue culture; Diagnostic Test: Next Generation Sequencing
- Septic (infected) Revision Spine Surgery: Spine surgery for known infection specifically: epidural abscess or septic revision. Epidural abscess must be managed surgically for inclusion. Septic revision cases include any surgery to address infected hardware from a previous spinal surgery.
  Interventions: Diagnostic Test: Tissue culture; Diagnostic Test: Next Generation Sequencing

INTERVENTIONS:
Diagnostic Test: Tissue culture — Discarded tissue collected during surgery will be sent to the hospital microbiological lab for aerobic and anaerobic
Diagnostic Test: Next Generation Sequencing — Discarded tissue collected during surgery will be sent to an outside lab for testing using next generation sequencing (NGS)

SUMMARY:
During revision spinal surgery for aseptic indications, there remains a concern that the failure may have resulted from undetectable subclinical infection. In the common revision indications of hardware loosening and adjacent segment disease it is possible that bacterial colonization and low-grade infection precipitated the failure event. There is also significant controversy on the role infectious processes have in the development of degenerative disc disease (modic changes). In particular, this study will investigate whether discogenic colonization with Propionibacterium acnes (P. acnes) can be associated with modic changes. Whereas, in surgery for known spinal infection, epidural abscess and septic revisions, it is possible that standard culture techniques fail to detect polymicrobial flora or accurate speciation. This may lead to inappropriate antibiotic management that is not addressing the range of pathology present. There remains an incomplete understanding of the role that subclinical infection plays in aseptic spinal revision surgery and degenerative disc disease

ELIGIBILITY:
Inclusion Criteria:

* All patients >18 years of age undergoing spinal surgery

Exclusion Criteria:

* All patients <18 years of age undergoing spinal surgery

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who are having spine surgery who are >18 years old for degenerative disease, infection, and malignancy.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2021-02-18 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | 1 year
  complications that patients experience after surgery will be noted from the patient chart after they have been evaluated by their surgeon
Patient Satisfaction | 1 year
  will be measured using the Short Form 12 Physical and Mental Score (SF-12)
Patient pain | 1 year
  will be measured using the Visual Analog Scale Neck and Arm Pain Score (VAS)

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States